CLINICAL TRIAL: NCT01778309
Title: Effects of NAC Supplementation on Skeletal Muscle Performance Following Aseptic Injury Induced by Exercise
Brief Title: NAC Supplementation and Skeletal Muscle Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Assistant Professor, Democritus University of Thrace
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: NACEXERCISE2011; CE-80739 (Other: Tzelalis Sports Medicine co.)
Record Dates: First submitted 2013-01-21; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Skeletal Muscle Damage; Skeletal Muscle Performance; Intgracellular Signaling in Skeletal Muscle; Inflammatory Status
Keywords: aseptic inflammation; skeletal muscle function; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- n-acetylcysteine/placebo supplementation (Experimental): n-acetylcysteine supplementation, orally in three daily dosages, at 20 mg/kg/day, daily for eight days after exercise placebo, orally in three daily dosages, content: 500 mL drink that contained water (375 mL), sugar-free cordial (125 ml), and 2 g of low-calorie glucose/dextrose powder.
  Interventions: Dietary Supplement: n-acetylcysteine supplementation

INTERVENTIONS:
Dietary Supplement: n-acetylcysteine supplementation — n-acetylcysteine administration: 20 mg//kg/day, orally, daily for eight days following exercise
  placebo administration: 500 mL orally, daily for eight days following exercise
  Other Names: Exercise-induced skeletal muscle damage

SUMMARY:
In this investigation the investigators utilized NAC administration to foster GSH availability during an 8-day period following eccentric exercise-induced muscle damage in order to test our hypotheses: i) antioxidant supplementation does not disturb performance and adaptations induced by exercise-induced muscle injury and ii) redox status perturbations in skeletal muscle are pivotal for the regulation of muscle' inflammatory response and repair.

DETAILED DESCRIPTION:
The major thiol-disulfide couple of reduced (GSH) and oxidized glutathione (GSSG) is a key-regulator of major transcriptional pathways regulating aseptic inflammation and recovery of skeletal muscle following aseptic injury. Antioxidant supplementation may hamper exercise-induced cellular adaptations.

Our objective was to examine how thiol-based antioxidant supplementation affects skeletal muscle's performance and redox-sensitive signalling during the inflammatory and repair phases associated with exercise-induced micro-trauma.In a double-blind, counterbalanced design, 12 men received placebo (PLA) or N-acetylcysteine (NAC, 20 mg/kg/day) following muscle-damaging exercise (300 eccentric contractions). In each trial, muscle performance was measured at baseline, post-exercise, 2h post-exercise and daily for 8 consecutive days. Muscle biopsies from vastus lateralis and blood samples were collected pre-exercise and 2h, 2d, and 8d post-exercise.

ELIGIBILITY:
Inclusion Criteria:

a) recreationally trained as evidenced by their maximal oxygen consumption levels (VO2max >45 ml/kg/min), b) were engaged in systematic exercise at least three times/week for ≥12 months), c) non-smokers, d) abstained from any vigorous physical activity during the study, e)abstained from consumption of caffeine, alcohol, performance-enhancing or antioxidant supplements, and medications during the study.

Exclusion Criteria:

a) a known NAC intolerance or allergy, b) a recent febrile illness, c) history of muscle lesion, d) lower limb trauma

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in reduced glutathione in blood | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
  Concentration of reduced glutathione in red blood cells
Change in reduced glutathione in muscle | one hour before exercise, 2 hours post-exercise, 2 days post-exercise, 8 days post-exercise
  concentration of reduced glutathione in quadriceps skeletal muscle group
Change in protein carbonyls in red blood cells and serum | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
  concentration of protein carbonyls
Change in protein carbonyls in muscle | one hour before exercise, 2 hours post-exercise, 2 days post-exercise, 8 days post-exercise
  protein carbonyl concentration in vastus lateralis skeletal muscle
Change in thiobarbituric acid reactive substances in red blood cells and serum | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
  thiobarbituric acid reactive substances concentration in serum and red blood cells
Change in thiobarbituric acid reactive substances in muscle | one hour before exercise, 2 hours post-exercise, 2 days post-exercise, 8 days post-exercise
  thiobarbituric acid reactive substances concentration in vastus lateralis skeletal muscle
Change in oxidized glutathione in red blood cells and blood | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
  Concentration of oxidized glutathione in red blood cells and whole blood
Change in total antioxidant capacity in serum | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in oxidized glutathione in muscle | one hour before exercise, 2 hours post-exercise, 2 days post-exercise, 8 days post-exercise
  concentration of oxidized glutathione in vastus lateralis skeletal muscle
Change in catalase activity in red blood cells and serum | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in glutathione peroxidase activity in red blood cells | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in creatine kinase activity in plasma | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in C-reactive protein in plasma | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in macrophage infiltration in muscle | one hour before exercise, 2 hours post-exercise, 2 days post-exercise, 8 days post-exercise
Change in white blood cell count in blood | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in neutrophil count in blood | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in fatty acid binding protein in plasma | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in cortisol concentration in blood | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in testosterone concentration in plasma | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
Change in cytokine concentration in plasma | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
  Measurement of IL-1β, IL-4, IL-6, TNF-α, IL-8, IL-10, IL-12p70 concentrations in plasma
Change in adhesion molecule concentration in blood | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
  Measurement of ICAM-1, VCAM-1, sP-selectin, sE-selectin concentrations in plasma
Change in intracellular signalling proteins in muscle | one hour before exercise, 2 hours post-exercise, 2 days post-exercise, 8 days post-exercise
  Measurement of phosphorylation levels of protein kinase B (Akt), mammalian target of rapamycin (mTOR), serine/threonine kinase (p70S6K), ribosomal protein S6 (rpS6), nuclear factor κB (NFκB), serine⁄threonine mitogen activated protein kinase (p38-MAPK) in vastus lateralis muscle.
Change in myogenic determination factor (MyoD) protein levels in muscle | one hour before exercise, 2 hours post-exercise, 2 days post-exercise, 8 days post-exercise
  MyoD expression in vastus lateralis muscle
Change in tumor necrosis factor α in muscle | one hour before exercise, 2 hours post-exercise, 2 days post-exercise, 8 days post-exercise
  Protein levels of TNF-α in vastus lateralis muscle

SECONDARY OUTCOMES:
Change in muscle function of knee extensor and flexor muscle | one hour before exercise, 5 minutes post-exercise, 2 hours post-exercise, daily for 8 days post-exercise
  assessment of muscle peak and mean torque of knee extensors and flexors on an isokinetic dynamometer at 0, 90 and 180 degrees/sec
Body composition | One day before exercise
  Assessment of percent (%) lean body mass.
Maximal aerobic capacity | One day before exercise
  Assessment of maximal oxygen consumption, an indice of cardiovascular conditioning
Change in profile of dietary intake | one hour before exercise, daily for 8 days post-exercise
  Assessment of dietary intake with emphasis on antioxidant element intake
Change in side effect occurence | one hour before exercise, daily for 8 days post-exercise
  The prevalence of potential side-effects (such as headaches or abdominal pain or any other discomfort) was monitored using a subjective 0-10 side-effects scale on a daily bases by an unblinded investigator (for ethical reasons).

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis F Fatouros, Ph.D., Principal Investigator — Democritus University of Thrace, Greece
Locations (1):
- Laboratory of Physical Education & Sport Performance, Komotini, Thrace, Greece

REFERENCES:
- [Derived] Michailidis Y, Karagounis LG, Terzis G, Jamurtas AZ, Spengos K, Tsoukas D, Chatzinikolaou A, Mandalidis D, Stefanetti RJ, Papassotiriou I, Athanasopoulos S, Hawley JA, Russell AP, Fatouros IG. Thiol-based antioxidant supplementation alters human skeletal muscle signaling and attenuates its inflammatory response and recovery after intense eccentric exercise. Am J Clin Nutr. 2013 Jul;98(1):233-45. doi: 10.3945/ajcn.112.049163. Epub 2013 May 29. PMID 23719546